CLINICAL TRIAL: NCT01873144
Title: High Flow Therapy vs Hypertonic Saline in Bronchiolitis Treatment. Randomized Controlled Trial
Brief Title: High Flow Therapy vs Hypertonic Saline in Bronchiolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Spain (Other Government)
Responsible Party: Principal Investigator, MªMercedes Bueno Campaña, Dr, Ministry of Health, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC11-437
Record Dates: First submitted 2013-05-29; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Acute Viral Bronchiolitis
Keywords: Bronchiolitis; Hypertonic saline solution; High-flow oxygen therapy; Respiratory distress; Comfort
MeSH Terms: conditions — Bronchiolitis; Dyspnea | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HSS (3%) + epinephrine (Active Comparator): Nebulized solution containing 0.5 mL/kg (maximum 3 mL) of epinephrine 1/1000 plus 2 mL of HSS(3%) every 4h for three times and afterwards at physician in charge criteria.
  Interventions: Drug: Epinephrine 1/1000; Drug: HSS 3%
- HHHFNC+epinephrine+Normal Saline(0.9%) (Experimental): Flow depending on weight (Tidal volume x respiratory rate x 9) and nebulized solution containing 0.5 mL/kg (maximum 3 mL) of epinephrine 1/1000 plus 2 mL of Normal Saline (NS) (0.9%) every 4h and afterwards at physician in charge criteria.
  Interventions: Drug: Epinephrine 1/1000; Device: HHHFNC; Drug: NS (0.9%)

INTERVENTIONS:
Drug: Epinephrine 1/1000 — Nebulization of 0.5 mL/kg (maximum 3 mL) of epinephrine 1/1000 every 4h for three times and afterwards at physician in charge criteria
  Other Names: Adrenaline 1/1000; Adrenalin 1/1000
Drug: HSS 3% — Nebulization 2 mL of HSS (3%)+ epinephrine every 4h for three times and afterwards at physician in charge criteria
  Arms: HSS (3%) + epinephrine
Device: HHHFNC — Precision Flow (Vapotherm Inc. Stevensville, Maryland, US ) and RT329 (Fisher and Paykel Healthcare, Auckland, New Zealand) were the dispositive used depending on the availability. Fisher and Paykel nasal cannula was used in both devices, depending on age
  Arms: HHHFNC+epinephrine+Normal Saline(0.9%)
Drug: NS (0.9%) — Nebulization of 2 mL of NS (0.9%)+ epinephrine every 4h for three times and afterwards at physician in charge criteria
  Other Names: Normal saline solution 0.9%; Physiologic saline solution
  Arms: HHHFNC+epinephrine+Normal Saline(0.9%)

SUMMARY:
The purpose of this study is to demonstrate that heated, humidified, high-flow nasal cannula (HHHFNC) is superior to hypertonic saline solution (HSS) in the treatment of moderate acute viral bronchiolitis in infants in improving respiratory distress and comfort and reducing length of hospital stay (LOS) and admission to Pediatric Intensive Care Unit (PICU).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months or less
* Moderate (Respiratory Distress Assessment Instrument score of 4 or greater) viral bronchiolitis (as defined by McConnockie)
* Meeting Admission criteria

Exclusion Criteria:

* History of prematurity
* Chronic lung disease
* Cystic fibrosis
* Congenital heart disease
* Neuromuscular disease
* Airway anomalies
* Immunodeficiency
* Those requiring immediate intubation and ventilation.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Difference in mean Respiratory Assessment Change Score (RACS) between groups in every time considered | Every 4h for three consecutive times beginning in the moment of inclusion in the study and after every 8h for three consecutive times (average of 36h)
  RACS is calculated by combining 2 values: the difference between the Respiratory Distress Assessment Instrument (RDAI) score before and after treatment, plus a value of +1 for each 10% improvement (decrease) in the posttreatment respiratory rate (RR) or a value of -1 for each 10% worsening (increase) in RR.

SECONDARY OUTCOMES:
Difference in mean comfort score along the monitoring period between groups | Every 8h for 6 consecutive times (two days) beginning in the moment of inclusion in the study
  A scale was used for comfort evaluation . It is based on 4 items: rest, feeding, alertness and facial expression (facial pictures).Minimum 4-Maximum 16

OTHER OUTCOMES:
Length of hospital stay (LOS) in days in both groups | Participants will be followed for the duration of hospital stay, an expected average of 5 days
Admission to Pediatric Intensive Care Unit PICU (rate) in both groups | Transfer to PICU at any time during hospitalization
  Transfer to PICU criteria were defined.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Bueno, MD, Principal Investigator — Department of Pediatrics and Neonatology. Hospital Universitario Fundacion Alcorcon. Madrid. SPAIN
Locations (2):
- Spain (2):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid

REFERENCES:
- [Derived] Bueno Campana M, Olivares Ortiz J, Notario Munoz C, Ruperez Lucas M, Fernandez Rincon A, Patino Hernandez O, Calvo Rey C. High flow therapy versus hypertonic saline in bronchiolitis: randomised controlled trial. Arch Dis Child. 2014 Jun;99(6):511-5. doi: 10.1136/archdischild-2013-305443. Epub 2014 Feb 12. PMID 24521787